CLINICAL TRIAL: NCT04795037
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Safety, Tolerability, and Pharmacokinetic Study of Escalating Single and Multiple Doses of CU06-1004 in Healthy Subjects
Brief Title: First-In-Human Study of CU06-1004 Following Single and Multiple Ascending Doses in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Curacle Co., Ltd. (Industry)
Collaborators: KCRN Research, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CU06-1004-DME-01
Record Dates: First submitted 2021-03-05; First posted 2021-03-12 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Diabetic Macular Edema
Keywords: DME; Endothelial dysfunction blocker
MeSH Terms: interventions — CU06-1004

STUDY DESIGN:
Intervention Model Description: A Single Ascending Dose(SAD) study with 7 Cohorts including 1 Cohorts for Food effect (FE) assessment with 8 subjects each (6 active and 2 placebo) and A Multiple Ascending Dose(MAD) study with 3 Cohorts with 8 subjects each (6 active and 2 placebo).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- CU06-1004 for SAD (Experimental): * Fifty-six (56) healthy subjects are planned to be enrolled in 7 cohorts
  * 6 of out 8 subjects per cohort will be randomized to receive CU06-1004
  Interventions: Drug: CU06-1004, Single dose
- Placebo for SAD (Placebo Comparator): * Fifty-six (56) healthy subjects are planned to be enrolled in 7 cohorts
  * 2 of out 8 subjects per cohort will be randomized to receive placebo
  Interventions: Drug: Placebo
- CU06-1004 for MAD (Experimental): * Twenty-four (24) healthy subjects are planned to be enrolled in 3 cohorts
  * 6 of out 8 subjects per cohort will be randomized to receive CU06-1004
  Interventions: Drug: CU06-1004, Multiple doses
- Placebo for MAD (Placebo Comparator): * Twenty-four (24) healthy subjects are planned to be enrolled in 3 cohorts
  * 2 of out 8 subjects per cohort will be randomized to receive placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CU06-1004, Single dose — Single dose of CU06-1004, 7 dose levels, oral capsule : 6 Cohorts (100mg, 300mg, 600mg, 900mg, 1200mg, 300mg bid) + 1 Cohort (Food effect)＊
  ＊Cohort S7(TBD mg) will receive a single oral dose of CU06-1004 or placebo under fed conditions. When administered under fed conditions, CU06-1004 or placebo will be administered following a high-fat/high-calorie breakfast. Cohort S7 will be conducted following completion of Cohort S5
  Other Names: SAC-1004; CU06; CU06-RE
  Arms: CU06-1004 for SAD
Drug: CU06-1004, Multiple doses — Multiple doses of CU06-1004, 7 days, 3 dose levels＊, oral capsule
  ＊The dose levels, regimen (i.e., schedule), and conditions (i.e., fasted versus fed conditions) will be determined based on the safety, tolerability, and plasma PK data from SAD
  Other Names: SAC-1004; CU06; CU06-RE
  Arms: CU06-1004 for MAD
Drug: Placebo — Placebo matched to CU06-1004, oral capsule
  Arms: Placebo for MAD; Placebo for SAD

SUMMARY:
This clinical trial is the first-in-human study of CU06-1004. The purpose of this phase 1 study is to assess the safety and tolerability of single and multiple ascending oral doses of CU06-1004 in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, adult, male or female (of non-childbearing potential only), 19-55 years of age, inclusive, at screening.
2. Body mass index (BMI) ≥ 18.0 and ≤ 32.0 kg/m2 at screening.
3. Continuous non-smoker who has not used nicotine-containing products for at least 3 months prior to the first dosing and throughout the study, based on subject self-reporting.
4. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs or ECGs, as deemed by the PI or designee.
5. Female must be of non-childbearing potential and must have undergone one of the following sterilization procedures at least 6 months prior to the first dosing:

   * hysteroscopic sterilization;
   * bilateral tubal ligation or bilateral salpingectomy;
   * hysterectomy;
   * bilateral oophorectomy; or be postmenopausal with amenorrhea for at least 1 year prior to the first dosing and follicle-stimulating hormone (FSH) serum levels consistent with postmenopausal status.
6. A non-vasectomized, male subject must agree to use a condom with spermicide or abstain from sexual intercourse during the study until 90 days after the last dosing.

   (No restrictions are required for a vasectomized male provided his vasectomy has been performed 4 months or more prior to the first dosing. A male who has been vasectomized less than 4 months prior to the first dosing must follow the same restrictions as a non-vasectomized male).
7. If male, must agree not to donate sperm from the first dosing until 90 days after the last dosing.
8. Able to swallow multiple capsules.
9. Understands the study procedures in the informed consent form (ICF), and be willing and able to comply with the protocol.

Exclusion Criteria:

1. Is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
2. History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI or designee.
3. History of any illness that, in the opinion of the PI or designee, might confound the results of the study or poses an additional risk to the subject by their participation in the study.
4. History or presence of alcohol or drug abuse within the past 2 years prior to the first dosing.
5. History or presence of hypersensitivity or idiosyncratic reaction to the study drug or related compounds.
6. Female subjects of childbearing potential.
7. Female subjects with a positive pregnancy test at screening or first check-in or who are lactating.
8. Positive urine drug or alcohol results at screening or first check-in.
9. Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV).
10. Seated blood pressure is less than 90/40 mmHg or greater than 140/90 mmHg, at screening.
11. Seated heart rate is lower than 40 bpm or higher than 99 bpm at screening.
12. QTcF interval is >460 msec (males) or >470 msec (females) or has ECG findings deemed abnormal with clinical significance by the PI or designee at screening.
13. Unable to refrain from or anticipates the use of:

    * Any drug, including prescription and non-prescription medications, herbal remedies, or vitamin supplements (especially sulforaphane-containing supplement) beginning 14 days prior to the first dosing and throughout the study. After randomization, acetaminophen (up to 2 g per 24 hours) may be administered at the discretion of the PI or designee.
    * Food and beverages containing xanthines/caffeine for 24 hours prior to the first dosing (small amounts of caffeine derived from normal foodstuffs e.g.,250 mL/8 oz./1 cup decaffeinated coffee or other decaffeinated beverage, per day, with the exception of espresso; 45 g/1.5 oz. chocolate bar, per day, would not be considered a deviation to this restriction).
    * Food and beverages containing alcohol for 48 hours prior to the first dosing.
    * Food and beverages containing grapefruit/Seville orange for 14 days prior to the first dosing.
    * Food and beverages containing vegetables from the mustard green family (e.g., kale, broccoli, watercress, collard greens, kohlrabi, Brussels sprouts, mustard) and charbroiled meats for 14 days prior to the first dosing.
14. Has received COVID-19 vaccine within 30 days of first dosing and until the end of the study.
15. Has been on a diet incompatible with the on-study diet, in the opinion of the PI or designee, within the 30 days prior to the first dosing and throughout the study.
16. Is lactose intolerant (FE cohort only).
17. Donation of blood or significant blood loss within 56 days prior to the first dosing.
18. Plasma donation within 7 days prior to the first dosing.
19. Participation in another clinical study within 30 days prior to the first dosing. The 30-day window will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to the first dose of study drug in the current study.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2022-06-25 (Actual)

PRIMARY OUTCOMES:
The number and severity of treatment emergent adverse events (TEAEs) | From the date of first dose through 7 days after the last dose
  To assess the safety and tolerability of single and multiple ascending oral doses of CU06-1004 in healthy adult subjects.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | Day 1 through Day 4 (SAD), Day 1 through Day 10 (MAD)
  To assess Cmax of single and multiple ascending oral doses of CU06-1004 in healthy adult subjects
Time to reach maximum plasma concentration (Tmax) | Day 1 through Day 4 (SAD), Day 1 through Day 10 (MAD)
  To assess Tmax of single and multiple ascending oral doses of CU06-1004 in healthy adult subjects
Area under the concentration-time curve (AUC) | Day 1 through Day 4 (SAD), Day 1 through Day 10 (MAD)
  To assess AUC of single and multiple ascending oral doses of CU06-1004 in healthy adult subjects
Terminal elimination rate constant (Kel) | Day 1 through Day 4 (SAD), Day 1 through Day 10 (MAD)
  To assess Kel of single and multiple ascending oral doses of CU06-1004 in healthy adult subjects
Terminal elimination half-life (t½) | Day 1 through Day 4 (SAD), Day 1 through Day 10 (MAD)
  To assess t½ of single and multiple ascending oral doses of CU06-1004 in healthy adult subjects
Maximum plasma concentration (Cmax) under fed conditions | Day 1 through Day 4 (SAD)
  To assess Cmax of single oral dose under fed conditions
Area under the concentration-time curve (AUC) under fed conditions | Day 1 through Day 4 (SAD)
  To assess AUC of single oral dose under fed conditions
Amount of unchanged drug excreted in the urine collection (Ae) | Day 1 through Day 4 (SAD), Day 1 through Day 10 (MAD)
  To assess Ae of single and multiple ascending oral doses of CU06-1004 in healthy adult subjects
Renal Clearance (CLR) | Day 1 through Day 4 (SAD), Day 1 through Day 10 (MAD)
  To assess CLR of single and multiple ascending oral doses of CU06-1004 in healthy adult subjects
Fraction of drug excreted unchanged in urine (Fe) | Day 1 through Day 4 (SAD), Day 1 through Day 10 (MAD)
  To assess Fe of single and multiple ascending oral doses of CU06-1004 in healthy adult subjects

CONTACTS AND LOCATIONS:
Overall Officials: Ji-Hye Kang, Ph.D, Study Director — Curacle Co., Ltd.
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maganti L, Panebianco DL, Maes AL. Evaluation of methods for estimating time to steady state with examples from phase 1 studies. AAPS J. 2008;10(1):141-7. doi: 10.1208/s12248-008-9014-y. Epub 2008 Feb 28. PMID 18446514
- [Background] Schuirmann DJ. A comparison of the two one-sided tests procedure and the power approach for assessing the equivalence of average bioavailability. J Pharmacokinet Biopharm. 1987 Dec;15(6):657-80. doi: 10.1007/BF01068419. PMID 3450848